CLINICAL TRIAL: NCT07160621
Title: Culturally Adapted Mobile Treatment of Chronic Pain in Adolescent Survivors of Pediatric Cancer: A Randomized Clinical Trial
Acronym: ADAPTED2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ADAPTED2; NCI-2025-06050 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Childhood Cancer Survivor; Chronic Pain
Keywords: Adult Caregiver; Adolescent Survivor
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy; Educational Status; Patient Education as Topic; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (mobile CBT) (Experimental): Participants who are randomized to receive mobile CBT for chronic pain.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Other: Questionnaires
- Arm II (Patient education) (Sham Comparator): Participants who are randomized to receive educational materials about chronic pain.
  Interventions: Behavioral: Education; Other: Questionnaires

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Receive mobile CBT
  Other Names: CBT, CBT, cognitive behavior therapy, cognitive therapy, CT
  Arms: Arm I (mobile CBT)
Behavioral: Education — Receive educational materials
  Other Names: Psychoeducation; patient education
  Arms: Arm II (Patient education)
Other: Questionnaires — Ancillary studies

SUMMARY:
The purpose of the study is to determine if an adapted mobile cognitive behavioral therapy (CBT) app (WebMAP Onc) is more effective than standard pain education in reducing chronic pain and improving daily functioning in adolescent survivors of pediatric cancer.

This randomized study led by St. Jude Children's Research Hospital will involve 204 participants (102 adolescent survivors and 102 caregivers) across four U.S. hospitals. Outcomes include pain reduction, improved function, and the role of social determinants of health. Assessments occur at baseline, post-treatment, and 3-month follow-up.

DETAILED DESCRIPTION:
Survivors of childhood cancer with lasting pain may have problems with daily life, such as paying attention, sleeping, or daily activities. A mobile cognitive behavioral therapy program (App) and patient education materials may be helpful for survivors with pain. Researchers at St. Jude Children's Research Hospital want to see if these tools can used to improve pain in survivors. Participants will be recruited from 4 sites: St. Jude Children's Research Hospital (SJCRH), Children's Healthcare of Atlanta (CHOA), Texas Children's Hospital (TCH), and Seattle Children's Hospital (SCH).

Standard treatment for pain that continues after cancer and its treatment may include pain education, medication and/or cognitive behavioral therapy. Cognitive behavioral therapy (CBT) is a treatment that focuses on helping people change how they think and feel about pain. This treatment is often delivered in person.

Participants will be asked to either use a mobile CBT program or review educational materials about pain for 6 weeks. For those using the CBT program, the program can be accessed at their convenience through an App on their phone and they will be asked to use the App at least 2 to 3 days per week.

Primary Objective:

To conduct a randomized clinical trial to determine the efficacy of adapted mobile CBT vs. patient education to improve pain intensity and functional disability post-intervention in a racially/ethnically and geographically diverse sample of adolescent survivors of childhood cancer with chronic pain.

Secondary Objective:

To investigate longitudinal associations between patient-reported comorbidities including symptoms of depression, anxiety, sleep quality, fatigue, physical functioning, and pain medication use with changes in pain intensity and functional disability.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent Participants

  * 10-17-year-old survivors of childhood cancer or those who received cancer directed therapies (e.g., Langerhan's Histiocytosis)
  * At least one-year post treatment completion
  * Pain present for 3 months or longer
  * Pain interfering with at least one area of daily functioning
* Parent/Caregiver Participants

  * ≥ 18 years of age
  * Legally authorized to provide informed consent for the adolescent participant

Exclusion Criteria:

* Adolescent Participants

  * Serious comorbid psychiatric condition
  * Current substance abuse as determined by the Substance Use Screening Questionnaire
  * History of development delay or significant cognitive impairment

    * Note: A participant who completed the feasibility study (ADAPTED) cannot participate in the subsequent clinical trial (ADAPTED2)
* Parent/Caregiver Participants

  * Not fluent in English or Spanish
  * Unable to provide consent for own participation or for the participation of the adolescent participant

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Up to 8 weeks from start of study
  The Brief Pain Inventory-Short Form (BPI) includes a 4-item pain severity scale. Participants rate their worst and least pain in the last 24 hours, average pain, and current pain. This measure includes a body diagram to allow participants to indicate where they experience the most pain and has a 10-point rating scale (No Pain to Pain As Bad As You Can Imagine). The higher scores indicate greater pain. The Brief Pain Inventory pain intensity has good internal consistency in survivors of childhood cancer (α=0.87).
Pain interference | Up to 8 weeks from start of study
  The Functional Disability Inventory (FDI) is a 15-item measure assessing difficulty performing daily activities in home, school, and social domains with higher scores indicating greater pain-related disability. The measure has a 4-point rating scale (No Trouble to Impossible) for performing daily activities. The Functional Disability Inventory has good internal consistency (α=0.85-0.92) and test-retest reliability (r=0.48-0.80).
Pain catastrophizing | Up to 8 weeks from start of study
  The Pain Catastrophizing Scale, Child version (PCS-C) is a 13-item self-report measure of overly negative attitudes of pain and it consists of three scales of rumination, magnification and helplessness. The 5-point rating scale (Not at All to Extremely). Higher scores indicate more pain catastrophizing. This measure has good reliability (Cronbach's α=0.90) in a clinical sample of children and adolescents with chronic or recurrent pain.
Depression | Up to 8 weeks from start of study
  The PROMIS Pediatric Depressive Symptoms is an 8-item measure of self-reported symptoms of low mood in children and adolescents over the past 7 days. The measure has a 5-point rating scale (Never to Almost Never). Higher scores indicate greater symptoms.
Anxiety | Up to 8 weeks from start of study
  The PROMIS Pediatric Anxiety is an 8-item measure of self-reported symptoms of anxiety symptoms in children and adolescents over the past 7 days. The measure has a 5-point rating scale (Never to Almost Always). Higher scores indicate greater symptoms.
Cancer-related worry | Up to 8 weeks from start of study
  The Fear of Cancer Recurrence Inventory is a 9-item measure developed specifically for survivors of childhood cancer (8-18 years) to assess the presence of fear of recurrence and perceived risk recurrence. The measure has 5-point rating scale (Not at All to A Great Deal). Higher scores indicate greater cancer-related worry. Internal consistency is good (ICC=0.88).
Physical functioning | Up to 8 weeks from start of study
  The PROMIS Pediatric Mobility is an 8-item measure of self-reported ability at physical activities in children and adolescents in the past 7 days. The measure has a 5-point rating scale (No Trouble to Not Able to Do). Higher scores indicate greater ability. It has excellent test-retest reliability (ICC=0.73) and adequate internal consistency (Cronbach's α=0.73-0.74). The PROMIS Pediatric Upper Extremity is an 8-item measure of self-upper extremity function in the past 7 days with higher score indicating greater ability. It has excellent test-retest reliability (ICC=0.71) and adequate internal consistency (Cronbach's α=0.62-0.63). Both measures are sensitive to change in participants with chronic pain.
Peer relations | Up to 8 weeks from start of study
  The PROMIS Pediatric Peer Relationship is an 8-item measure that assesses the quality of peer relationships. The measure has a 5-point rating scale (Never to Almost Always). Higher score indicating higher quality. It has excellent test-retest reliability (ICC=0.81) and excellent internal consistency (Cronbach's α=0.83-0.84).
Fatigue | Up to 8 weeks from start of study
  The PROMIS Pediatric Fatigue is a 10-item measure that assesses symptoms of fatigue in the past 7 days. The measure has a 5-point rating scale. Higher scores indicate more fatigue. It has excellent test-retest reliability (ICC=0.76) and internal consistency (Cronbach's α=0.87).
Sleep | Up to 8 weeks from start of study
  The Adolescent Sleep Wake Scale (ASWS) short form93 is a 10-item measure of behavioral sleep patterns in adolescents. The measure is a 6-point rating scale (Never to Always). Higher scores indicate better success of sleep quality. Internal consistency was good (α=0.74-0.84) in a pooled clinical sample of adolescents with mixed health conditions).93 Acceptable reliability was reported in a sample of ethnically diverse adolescents from an economically disadvantage community (α=0.70-0.90).94 We also will use the PROMIS Sleep-Related Impairment95 8-item measure to allow for assessment of sleep quality during the night as well as the impact of sleepiness on daytime function. This measure is validated for children and adolescents and assess sleep-related impairment over the past 7 days.
Opioid Use | Up to 8 weeks from start of study
  At each timepoint participants and/or their parents will be asked to list the names of their medications, doses taken, and the frequency with which the medications were taken over the past 2 weeks. Medications will be classified as anti-inflammatory (e.g., nonsteroidal anti-inflammatory drugs); regular (daily) opioids, opioid medication as required (PRN), adjuvant pain medications (e.g., anticonvulsants). Opioid doses will be converted to morphine equivalent doses (MED) using an opioid equivalence table.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Brinkman, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States